CLINICAL TRIAL: NCT06486727
Title: Efficacy and Safety of 675-nm Laser for Dorsal Hand Rejuvenation in Thai Patients
Brief Title: Efficacy and Safety of 675-nm Laser for Dorsal Hand Rejuvenation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Prof. Dr., Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Si 488/2024
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 675-nm laser (RedTouch) (Experimental): Paramete: Moveo, power 5 W, Energy/DOT 500 mJ/DOT then Standard, power 4 W, spacing 2000 μm, 1 pass per side for 4 times with 4-week interval
  Interventions: Device: Redtouch

INTERVENTIONS:
Device: Redtouch — 675-nm laser

SUMMARY:
This study aimed to evaluate efficacy and safety of 675-nm laser for dorsal hand rejuvenation in Thai patients. Twenty-six subjects aged 50 to 65 years diagnosed with wrinkle and solar lentigines on both dorsums of hands were included and treated with RedTouch for 3 times every 4 weeks. Then, they were follow up at 3 and 6 months after the final treatment. The measurement of 5-point Global Aesthetic Improvement Scale scores by physicians and subjects were conducted. Moreover, pigmentation level, wrinkle and texture were also recored using Antera. Elasticity was measured using Cutometer.

DETAILED DESCRIPTION:
RedTouch parameter included Moveo, power 5 W, Energy/DOT 500 mJ/DOT, then Standard, power 4 W, spacing 2000 μm, 1 pass per side.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with wrinkles and solar lentigines on both dorsum of hands

Exclusion Criteria:

* Pregnant or lactation
* Sugjects with a history of allergy to near-infrared wavelength or photosensitizing agents
* Subjects who have been treated with any kind of energy-based device on both dorsum of hands 6 months prior to the inclusion
* Subjects who have been injected with filler, or platelet-rich plasma on both dorsum of hands on their faces 6 months prior to the inclusion
* Active skin infections
* History of hypertrophic scars or keloids

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The change in pigmentation level, wrinkle and texture | Baseline, 4, 8, 12 weeks after the first treatment and 3, 6 months after the last treatment
  Using Antera®

SECONDARY OUTCOMES:
The change in elasticity | Baseline, 4, 8, 12 weeks after the first treatment and 3, 6 months after the last treatment
  Using Cutometer®
Overall improvement by physicians and patients | 4, 8, 12 weeks after the first treatment and 3, 6 months after the last treatment
  5-point GAIS
Adverse events | 4, 8, 12 weeks after the first treatment and 3, 6 months after the last treatment
  Side effects
Pain score | Baseline, 4, 8, 12 weeks after the first treatment
  Visual analog scale (0-10; no pain-worst pain possible)

CONTACTS AND LOCATIONS:
Overall Officials: Woraphong Manuskiatti, MD, Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: No